CLINICAL TRIAL: NCT01252225
Title: Effect of Lidocaine and Its Delivery in Patients With Chronic Cough
Brief Title: Lidocaine: Effect of Lidocaine in Chronic Cough
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Lidocaine1
Record Dates: First submitted 2010-11-29; First posted 2010-12-02 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Chronic Cough
Keywords: Chronic Cough; Lidocaine
MeSH Terms: conditions — Chronic Cough | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nebulised Lidocaine followed by Placebo throat spray (Active Comparator)
  Interventions: Drug: 10 % Lidocaine
- Nebulised Placebo followoed by Lidocaine Throat Spray (Active Comparator)
  Interventions: Drug: 10 % Lidocaine
- Nebulised placebo followed by placebo throat spray (Placebo Comparator)
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: 10 % Lidocaine — 600 mg Nebulised Lidocaine ( 6 mls of 10 % Lidocaine) one-off dose
  Other Names: Lidocaine; Lignocaine
  Arms: Nebulised Lidocaine followed by Placebo throat spray
Drug: 10 % Lidocaine — 100 mg Lidocaine ( 1 ml of 10 % Lidocaine) given as one-off throat spray.
  Other Names: Lidocaine; Lignocaine
  Arms: Nebulised Placebo followoed by Lidocaine Throat Spray
Drug: 0.9% saline — 6 mls of 0.9% saline nebulised followed by 1 ml of 0.9% saline as throat spray
  Arms: Nebulised placebo followed by placebo throat spray

SUMMARY:
People cough in order to clear their airways. Most coughs are caused by viruses and settle down by themselves, but some people develop persistent coughing which can be anywhere from 8 weeks to several years. This is called chronic cough. People with chronic cough find the symptom distressing and it can have a major impact on their quality of life. Patients with chronic cough often report a sensation at the back of their throat which makes them feel an urge to cough. There is some evidence that Lidocaine (an anaesthetic used during medical procedures) can suppress a person's cough when given to patients via a nebuliser (a machine that turns liquid into a fine mist).

It is currently unknown whether using a local anaesthetic, such as Lidocaine, in the form of a throat spray would successfully suppress a person's cough. A throat spray would be an easier treatment option in chronic cough patients. Thus, the investigators research aims to compare cough rates, severity and urge to cough scores between Lidocaine throat spray and nebulised Lidocaine.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, age 18 years and over.
* History of cough for more than 8 weeks.
* Normal chest x ray
* Chronic idiopathic cough or chronic cough resistant to treatment of specific triggers.

Exclusion Criteria:

* Smoking status:

  * Current smokers
  * Ex smokers with history of smoking > 20 pack years or those who have given up < 6 months ago.
* Prohibited medications:

  * Use of medications likely to suppress / affect cough including codeine, morphine, pregabalin, gabapentin, amitriptylline, angiotensin converting enzyme inhibitors (type 1) and baclofen.
  * Use of any anti-arrhythmic medication.
  * Use of cimetidine, beta blockers, or diuretics.
* Cardiovascular conditions:

  * Sinoatrial disease, bradycardia or all types of heart blocks.
  * History of ischaemic heart disease or heart failure.
  * Clinically significant abnormal electrocardiogram (ECG) at Screening or Baseline.
  * History of cardiac surgery
* Respiratory conditions:

  o Asthma.
* Central nervous system / Peripheral nervous system conditions:

  * Epilepsy.
  * Myasthenia gravis.
* Miscellaneous:

  * History of hepatic or renal dysfunction.
  * Porphyria
  * History of hypersensitivity to Lidocaine or related drugs.
  * Pregnancy or breast feeding.
  * Participation in another trial within the preceding 6 weeks.
  * Trauma or ulceration to oral mucosa.
  * History of chest or upper airway infection within the past 6 weeks.
  * Conditions which may affect cough response such as stroke, diabetes, Parkinson's Disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Objective cough counts over 10 hours post dose. Change in Urge to cough and Visual Analogue Score (VAS). | over 24 hours following treatment
  patients will wear a cough recorder device for a 24 hour period. The recordings will then be analysed to reveal how many times the patient coughed.

SECONDARY OUTCOMES:
Heart rate | over 2 hours
  to document any change in heart rate after treatment
Mouth Numbness | over 24 hours following treatment
  Duration of mouth numbness will be subjectively assessed by asking patients about the presence of mouth numbness and its duration after treatment.
Electrocardiogram (ECG) | 15 minutes after treatment
  ECG will be recorded before treatment and 15 minutes after treatment to rule out any arrhythmias

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Woodcock, MD, FRCP, Principal Investigator — University of Manchester
Locations (1):
- University Hospital of South Manchester, Manchester, United Kingdom